CLINICAL TRIAL: NCT03481725
Title: Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: A Non-Pharmacologic Alternative for the Treatment of Postoperative Pain
Brief Title: Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: A Department of Defense Funded Multicenter Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); Walter Reed National Military Medical Center (U.S. Federal Agency); Wake Forest University Health Sciences (Other); Augusta University (Other); The Cleveland Clinic (Other); Brooke Army Medical Center (U.S. Federal Agency); United States Naval Medical Center, San Diego (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); Womack Army Medical Center (U.S. Federal Agency); SPR Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pilot STIMULATION (DoD); NH170005 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Rotator Cuff Repair; Anterior Cruciate Ligament Reconstruction; Ankle Arthrodesis or Arthroplasty; Hallux Valgus Correction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Peripheral Nerve Stimulation (Experimental): ACTIVE percutaneous peripheral nerve stimulation with an ultrasound-guided percutaneous lead (SPR Therapeutics, Cleveland, Ohio) and wearable stimulator (SPR Therapeutics, Cleveland, Ohio) that generates electrical current
  Interventions: Device: ACTIVE peripheral nerve stimulation with a percutaneously inserted lead and wearable stimulator (SPR Therapeutics, Cleveland, Ohio)
- Sham (Sham Comparator): SHAM percutaneous peripheral nerve stimulation with an ultrasound-guided percutaneous lead (SPR Therapeutics, Cleveland, Ohio) and wearable stimulator (SPR Therapeutics, Cleveland, Ohio) that does NOT generate electrical current
  Interventions: Device: SHAM peripheral nerve stimulation with a percutaneously inserted lead and wearable SHAM stimulator (SPR Therapeutics, Cleveland, Ohio)

INTERVENTIONS:
Device: ACTIVE peripheral nerve stimulation with a percutaneously inserted lead and wearable stimulator (SPR Therapeutics, Cleveland, Ohio) — ACTIVE peripheral nerve stimulation with a percutaneously inserted lead and wearable stimulator (SPR Therapeutics, Cleveland, Ohio) that generates electric current for 14 days
  Arms: Peripheral Nerve Stimulation
Device: SHAM peripheral nerve stimulation with a percutaneously inserted lead and wearable SHAM stimulator (SPR Therapeutics, Cleveland, Ohio) — SHAM peripheral nerve stimulation with a percutaneously inserted lead and wearable stimulator (SPR Therapeutics, Cleveland, Ohio) that does not generate electric current for 14 days
  Arms: Sham

SUMMARY:
Postoperative pain is usually treated with opioids that have undesirable and sometimes dangerous side effects (e.g., vomiting and respiratory depression)-and yet over 80% of patients still experience inadequate pain relief. A novel, non-pharmacologic analgesic technique-percutaneous peripheral nerve stimulation (PNS)- holds extraordinary potential to greatly reduce or obviate opioid requirements and concurrently improve analgesia following painful surgery. This technique involves inserting an insulated electric lead adjacent to a target nerve through a needle prior to surgery using ultrasound guidance. Following surgery, a tiny electric current is delivered to the nerve resulting in potent pain control without any cognitive or adverse systemic side effects whatsoever. The electrical pulse generator (stimulator) is so small it is simply affixed to the patient's skin. The leads are already cleared by the US Food and Drug Administration to treat acute (postoperative) pain for up to 60 days; and, since percutaneous PNS may be provided on an outpatient basis, the technique holds the promise of providing potent analgesia outlasting the pain of surgery-in other words, the possibility of a painless, opioid-free recovery following surgery.

The current project is a multicenter, randomized, double-masked, placebo-controlled, parallel-arm clinical pilot study to (1) determine the feasibility and optimize the protocol of a planned definitive clinical trial; and (2) estimate the treatment effect of percutaneous PNS on pain and opioid consumption following moderate-to-severely painful ambulatory surgery compared with usual and customary opioid-based analgesia. This will allow determination of the required sample size for a subsequent definitive multicenter clinical trial. Combined, the pilot study and definitive trial have a strong potential to dramatically reduce or obviate postoperative opioid requirements and their resultant negative effects on both individuals and society; while concurrently improving analgesia, increasing the ability to function in daily life, decreasing the risk of transition from acute to chronic pain, and improving quality of life.

DETAILED DESCRIPTION:
This is a pilot or feasibility study (designated as UG3 by the Department of Defense) which will be a randomized, double-masked, placebo-controlled, parallel-arm, human subjects pilot study with two Specific Aims:

Specific Aim 1 (UG3): To determine the feasibility and optimize the protocol of the Implementation Phase (UH3) multicenter clinical trial that will compare percutaneous PNS with usual and customary opioid-based analgesia following moderate-to-severely painful ambulatory surgery.

Specific Aim 2 (UG3): To estimate the treatment effect of percutaneous PNS on pain and opioid consumption following moderate-to-severely painful ambulatory surgery compared with usual and customary opioid-based analgesia. This will allow determination of the required sample size of the definitive multicenter clinical trial of the Implementation Phase (UH3).

Anthropomorphic and demographic characteristics as well as baseline end points will be recorded/measured, including a pain score at the surgical site using the Numeric Rating Scale (NRS, 0-10), sensory deficits (measured with von Frey filaments within the cutaneous distribution of the target nerve), and muscle strength (measured with a pressure transducer).

Shoulder • Rotator cuff repair Brachial plexus trunks (lead & interscalene nerve block)

Knee • Anterior cruciate ligament repair with a patellar autograph Femoral lead & Adductor canal nerve block

Foot or ankle • Hallux valgus correction or Ankle arthrodesis/ arthroplasty Subgluteal sciatic lead and Popliteal sciatic nerve block

Insulated leads will be inserted prior to peripheral nerve block administration. The lead insertion sites will be cleansed with chlorhexidine gluconate and isopropyl alcohol, and a sterile, fenestrated drape applied. A portable ultrasound paired with either a linear or curved array transducer within a sterile sleeve will be used for lead insertion. The target nerve will be imaged in a transverse cross-sectional (short axis) view and a local anesthetic skin wheal raised lateral to the ultrasound transducer.

A needle and a pre-loaded, monopolar, helically-coiled, insulated lead (SPR Therapeutics, Cleveland, OH) will be inserted. Using an in-plane ultrasound approach, the needle tip will be advanced to the target nerve. The lead will be subsequently attached to an external stimulator (SPR Therapeutics). Accurate lead placement will be confirmed with subject reports of comfortable sensations over the surgical site without eliciting muscle contractions.

Stimulation parameters will be adjusted to improve stimulation coverage and comfort. Once optimum parameters have been determined, the needle will be withdrawn over the lead. The lead will be affixed to the skin with a sterile occlusive dressing. The stimulator will be set to deliver a range of currents. During their treatment, subjects can control these levels. Muscle strength will again be tested with the stimulator set for the optimal setting. The stimulator will be removed until after surgery.

Preoperatively, day of surgery. Subjects will continue to receive usual and customary local anesthetic-based analgesia. Because percutaneous PNS does not induce a sensory block and therefore does not provide anesthesia for the surgical procedure itself, we will continue to provide subjects with a preoperative single-injection local anesthetic-based peripheral nerve block (20 mL of ropivacaine 0.5% with epinephrine 1:400,000). In addition, surgeons will be permitted to infiltrate the surgical area with local anesthetic.

Treatment group assignment (randomization). Subjects will be allocated to a treatment only after confirmation of successfully-inserted electrical leads and surgical procedure initiation; and will be randomized to one of two possible treatment groups:

1. Current delivered via the electrical lead(s) [Experimental group]
2. No current delivered via the electrical lead(s) [Control group]

Randomization will be stratified by institution and anatomic lead location in a 1:1 ratio and in randomly chosen block sizes. Treatment group assignment will be conveyed to the enrolling sites via the same secure web-based system (RedCap) used to collect and collate all post-intervention endpoints. Stimulators are capable of programming to either (1) pass electrical current; or, (2) not pass electrical current. Importantly, these 2 modes (active and sham) are indistinguishable in appearance, and therefore investigators, subjects, and all clinical staff will be masked to treatment group assignment, with the only exception being the unmasked individual who programs the stimulator who will not have contact with the subject following randomization.

Subjects will be informed that often during postoperative active treatment with electrical current patients do not always have the sensations experienced during preoperative lead placement and once proper placement is confirmed with comfortable sensations, therapeutic levels of stimulation may be delivered sub-threshold (below the intensity required for sensation and still provide relief, which is factual/accurate). This protocol will ensure a randomized, double/triple-masked, sham/placebo-controlled trial. For the feasibility study (UG3), unmasking will occur 2 weeks following surgery to allow for protocol revisions, as necessary ("double masked" during initial data collection). In contrast, for the definitive pragmatic clinical trial (UH3) unmasking will not occur until statistical analysis for the entire investigation is complete (termed "triple masked").

Intraoperative course. The primary surgical anesthetic will be a general anesthetic, spinal anesthetic (bupivacaine) or exclusively the preoperative single-injection peripheral nerve block. Anesthetics that are also analgesics such as ketamine will not be used: the only permitted analgesic will be intravenous fentanyl, which will be minimal since all subjects will receive a single-injection peripheral nerve block immediately prior to surgery.

Postoperative course. Within the recovery room following surgery, the stimulators will be attached to the leads and activated, followed by end point assessment. Subjects who had a spinal anesthetic will have end points recorded following spinal resolution. Operating and recovery room pharmacologic analgesic requirements will be recorded.

Prior to discharge, subjects and their caretakers will be provided with verbal and written stimulator/lead instructions and the telephone and pager numbers of a local investigator available at all times. Subjects will be discharged home with their leads in situ. Subjects will be also be discharged with a prescription for an immediate-release oral opioid. Subjects will be contacted by telephone for end point collection (pain and analgesic consumption will be reported by phone on postoperative days 1, 2, 3, 4, 7, 11, and 15 as well as months 1 and 4). Lead removal will occur on postoperative day 14 (+/- 2 days) by healthcare providers. If the lead is removed following Day 14, the stimulator will be turned off on Day 14, and removed subsequently. Following study completion, the results will be mailed electronically or by the United States Postal Service to all enrolled subjects in written form using non-technical language.

Outcome measurements (end points). We have selected outcome measures that have established reliability and validity, with minimal inter-rater discordance, and are recommended for pain-related clinical trials by the World Health Organization and the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) consensus statement. Importantly, nearly all outcome measures are common data elements from the National Institute of Neurological Disorders and Stroke (NINDS). End points will be evaluated on postoperative days 0 (baseline), 1, 2, 3, 4, 7, 11, and 15 as well as months 1 and 4).

Demographic and medical history. Subjects will have demographic and anthropomorphic data collected based on NINDS case report form General Core and Demographics Modules and Guidelines, including age, sex, height, weight, educational level, employment status, marital status, and U.S. military service (e.g., none, discharged, active). In addition, the medical history based on the common data elements of the NINDS Medical, Family, Behavioral History, History of Disease/Injury Event, and Prior and Concomitant Medications Sub-Domains will be collected, and include the mechanism of original injury, medications (including analgesics), previous surgical procedures, comorbidities, existing sensory deficits of the target nerve distribution, preoperative pain levels measured on a Numeric Rating Scale for pain (including daily least, average, worst and current), and muscle strength if applicable (measured with a pressure transducer). In addition, since post-traumatic stress disorder (PTSD) may be associated with the severity of pain, at baseline we will apply the PTSD Checklist (PCL-C), a 20-item self-report measure reflecting symptoms of PTSD validated in military, Veteran, and civilian populations.

Data collection. Much of the surgical data from the day of surgery will be extracted from electronic health records to leverage data collection that occurs in health care delivery rather than requiring independent research data collection. Subject demographic, surgical and percutaneous PNS administration data will be uploaded from each enrolling center via the Internet to a secure, password-protected, encrypted central server (RedCap, Department of Outcomes Research, Cleveland Clinic, Cleveland, Ohio). All data collection following the day of enrollment (postoperative day 0)-regardless of enrolling center-will be collected by telephone from the University of California San Diego. Staff masked to treatment group assignment will perform all assessments.

UG3 Planning Phase Specific Aims. The investigation described above will accomplish the two Specific Aims of the UG3 Planning Phase:

Specific Aim 1 (UG3): To determine the feasibility and optimize the protocol of the Implementation Phase (UH3) multicenter clinical trial that will compare percutaneous PNS with usual and customary opioid-based analgesia following moderate-to-severely painful ambulatory surgery.

Specific Aim 2 (UG3): To estimate the treatment effect of percutaneous PNS on pain and opioid consumption following moderate-to-severely painful ambulatory surgery compared with usual and customary opioid-based analgesia. This will allow determination of the required sample size of the definitive multicenter clinical trial of the Implementation Phase (UH3).

** The primary end points will be cumulative opioid consumption and the mean value of the "average" daily surgical pain scores (measured with a Numeric Rating Scale) within the first 7 days following surgery (data collected Days 1, 2, 3, 4, and 7). In order to claim that percutaneous PNS is superior to usual and customary analgesia, at least one of Hypotheses 1 and 2 above must be superior while the other either superior or at least noninferior.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. undergoing one of the following surgical procedures: rotator cuff repair, anterior cruciate ligament repair with a patellar autograph, ankle arthrodesis or arthroplasty, hallux valgus correction
3. with a planned single-injection peripheral nerve block for postoperative analgesia

Exclusion Criteria:

1. chronic analgesic use including opioids (daily use within the 2 weeks prior to surgery and duration of use > 4 weeks)
2. neuro-muscular deficit of the target nerve(s)
3. compromised immune system based on medical history (e.g., immunosuppressive therapies such as chemotherapy, radiation, sepsis, infection), or other conditions that places the subject at increased risk
4. implanted spinal cord stimulator, cardiac pacemaker/defibrillator, deep brain stimulator, or other implantable neurostimulator whose stimulus current pathway may overlap
5. history of bleeding disorder
6. antiplatelet or anticoagulation therapies other than aspirin due to the risk of bleeding with a 20-gauge insertion needle
7. allergy to skin-contact materials (occlusive dressings, bandages, tape etc.)
8. incarceration
9. pregnancy
10. chronic pain of greater than 3 months of any severity in an anatomic location other than the surgical extremity
11. anxiety disorder
12. history of substance abuse
13. inability to contact the investigators during the treatment period, and vice versa (e.g., lack of telephone access).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-07-14 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2021-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University California San Diego
Locations (6):
- United States (6):
  - University California San Diego, San Diego, California
  - Naval Medical Center San Diego, San Diego, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Womack Army medical Center, Fort Bragg, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Brooke Army Medical Center, Fort Sam Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ilfeld BM, Gelfand H, Dhanjal S, Hackworth R, Plunkett A, Turan A, Vijjeswarapu AM, Cohen SP, Eisenach JC, Griffith S, Hanling S, Mascha EJ, Sessler DI. Ultrasound-Guided Percutaneous Peripheral Nerve Stimulation: A Pragmatic Effectiveness Trial of a Nonpharmacologic Alternative for the Treatment of Postoperative Pain. Pain Med. 2020 Dec 12;21(Suppl 2):S53-S61. doi: 10.1093/pm/pnaa332. PMID 33313729

RESULTS

PARTICIPANT FLOW:
Groups:
- Peripheral Nerve Stimulation: ACTIVE peripheral nerve stimulation with a percutaneously inserted lead and wearable stimulator that DOES generate electric current for 14 days
- Sham: SHAM peripheral nerve stimulation with a percutaneously inserted lead and wearable stimulator that does NOT generate electric current for 14 days
Period: Overall Study
Arm/Group | Peripheral Nerve Stimulation | Sham
Started | 31 | 34
Completed | 30 | 34
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peripheral Nerve Stimulation | Sham | Total
Number analyzed (Participants) | 31 | 34 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (16) | 55 (16) | 56 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 16 | 17 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 31 | 34 | 65
Height [Mean (Standard Deviation); unit: cm] | 172 (11) | 174 (10) | 173 (10)
Weight [Mean (Standard Deviation); unit: kg] | 80 (16) | 86 (20) | 83 (18)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27 (4) | 29 (5) | 28 (5)
Years of education [Mean (Standard Deviation); unit: years] | 17 (3) | 16 (3) | 17 (3)
Marital Status [Count of Participants; unit: Participants]
  Single | 9 | 9 | 18
  Currently Married | 18 | 23 | 41
  Others (separated and widowed) | 4 | 2 | 6
Military Status [Count of Participants; unit: Participants]
  Civilian (never in military) | 23 | 29 | 52
  Veteran | 8 | 3 | 11
  Active Duty | 0 | 2 | 2
Enrolling Center [Count of Participants; unit: Participants]
  Cedars-Sinai | 1 | 1 | 2
  University California San Diego | 28 | 28 | 56
  Naval Medical Center San Diego | 0 | 1 | 1
  Walter Reed National Military Medical Center | 1 | 2 | 3
  Womack Army Medical Center | 1 | 2 | 3
Surgical Procedure [Count of Participants; unit: Participants]
  Rotator cuff repair | 13 | 8 | 21
  Anterior cruciate ligament reconstruction | 1 | 3 | 4
  Ankle arthrodesis | 4 | 7 | 11
  Ankle arthroplasty | 4 | 5 | 9
  Hallux valgus | 9 | 11 | 20
Surgical side [Count of Participants; unit: Participants]
  Left | 10 | 19 | 29
  Right | 21 | 15 | 36
General anesthetic [Count of Participants; unit: Participants] | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption During First Postoperative Week
Description: Cumulative opioid dose from days 0-7, collected on days 0, 1, 2, 3, 4, and 7 for the previous 24 hours at each time point measured in morphine equivalents
Time Frame: Postoperative days 0-7
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Peripheral Nerve Stimulation | Sham
Number analyzed (Participants) | 31 | 34
mg | 5.0 [0 to 30.0] | 47.5 [25 to 90]

2. Primary Outcome: Average Pain During First Postoperative Week
Description: Mean value of the "average" pain scores measured using the numeric rating scale, collected on days 0, 1, 2, 3, 4, and 7 for the previous 24 hours at each time point. This is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain
Time Frame: Postoperative days 0-7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation | Sham
Number analyzed (Participants) | 31 | 34
score on a scale | 1.1 (1.1) | 3.1 (1.7)

3. Secondary Outcome: Opioid Consumption Individual Time Points
Description: Cumulative opioid dose of previous 24 hours (measured in morphine equivalents)
Time Frame: Postoperative days 1, 2, 3, 4, 7, 11, and 15; as well as Months 1 and 4
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Peripheral Nerve Stimulation | Sham
Number analyzed (Participants) | 31 | 34
mg
  Postoperative Day 1 | 0 [0 to 100] | 15 [0 to 20]
  Postoperative Day 2 | 5 [0 to 10] | 20 [10 to 30]
  Postoperative Day 3 | 0 [0 to 0] | 10 [0 to 20]
  Postoperative Day 4 | 0 [0 to 0] | 5 [0 to 20]
  Postoperative Day 7 | 0 [0 to 0] | 0 [0 to 10]
  Postoperative Day 11 | 0 [0 to 0] | 0 [0 to 5]
  Postoperative Day 15 | 0 [0 to 0] | 0 [0 to 0]
  Postoperative Month 1 | 0 [0 to 0] | 0 [0 to 0]
  Postoperative Month 4 | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Brief Pain Inventory, Short Form (Interference Domain)
Description: The Brief Pain Inventory (short form) interference domain is comprised of 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0 = no interference; 10 = complete interference]: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The score is calculated by adding the responses for each individual question resulting in a possible range of 0-70 (higher = worse).
Time Frame: Postoperative days 3, and 7; as well as Months 1 and 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peripheral Nerve Stimulation | Sham
Number analyzed (Participants) | 31 | 34
units on a scale
  Postoperative Day 3 | 2.6 (4.5) | 21.5 (17.9)
  Postoperative Day 7 | 2.5 (4.9) | 19.0 (17.0)
  Postoperative Month 1 | 4.0 (7.7) | 6.2 (10.4)
  Postoperative Month 4 | 1.6 (3.7) | 5.8 (12.3)

5. Secondary Outcome: Average Pain at Individual Time Points
Description: Mean of the "average" pain scores of previous 24 hours measured on a 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain
Time Frame: Postoperative days 1, 2, 3, 4, 7, 11, and 15; as well as Months 1 and 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation | Sham
Number analyzed (Participants) | 31 | 34
score on a scale
  Postoperative Day 1 | 1.8 (1.8) | 4.0 (2.6)
  Postoperative Day 2 | 1.3 (1.4) | 3.9 (2.1)
  Postoperative Day 3 | 0.9 (1.2) | 3.1 (2.3)
  Postoperative Day 4 | 0.7 (1.2) | 2.3 (2.0)
  Postoperative Day 7 | 0.6 (1.1) | 1.9 (2.1)
  Postoperative Day 11 | 0.3 (0.2) | 1.7 (1.4)
  Postoperative Day 15 | 0.9 (0.6) | 1.9 (1.6)
  Postoperative Month 1 | 0.5 (0.8) | 1.3 (1.8)
  Postoperative Month 4 | 0.3 (0.9) | 0.8 (1.7)

6. Secondary Outcome: Worst Pain at Individual Time Points
Description: Median of the worst pain scores of previous 24 hours measured on a 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain
Time Frame: Postoperative days 1, 2, 3, 4, 7, 11, and 15; as well as Months 1 and 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation | Sham
Number analyzed (Participants) | 31 | 34
score on a scale
  Postoperative Day 1 | 4 [0 to 6] | 7.8 [3 to 9]
  Postoperative Day 2 | 4 [2 to 6] | 7.5 [5 to 9]
  Postoperative Day 3 | 3 [0 to 4] | 6 [4 to 8]
  Postoperative Day 4 | 1.3 [0 to 4] | 4.3 [3 to 7]
  Postoperative Day 7 | 1.8 [0 to 3.5] | 3.5 [3 to 5]
  Postoperative Day 11 | 0.5 [0 to 2] | 3 [1 to 5]
  Postoperative Day 15 | 1.0 [0 to 5] | 2 [0 to 4.5]
  Postoperative Month 1 | 3.0 [0 to 4] | 2 [0 to 4]
  Postoperative Month 4 | 0 [0 to 1] | 1.5 [0 to 3]

7. Secondary Outcome: Least Pain at Individual Time Points
Description: Least pain scores of previous 24 hours measured on a 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain. Participants were asked "what was the lowest pain within the last 24 hours measured using the 0 to 10 scale, with 0 equal to no pain and 10 equal to the worst imaginable pain"?
Time Frame: Postoperative days 3 and 7; as well as Months 1 and 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation | Sham
Number analyzed (Participants) | 31 | 34
score on a scale
  Postoperative Day 3 | 0.2 (0.6) | 1.4 (1.8)
  Postoperative Day 7 | 0.2 (0.7) | 0.7 (1.6)
  Postoperative Month 1 | 0.1 (0.3) | 0.5 (1.0)
  Postoperative Month 4 | 0.3 (0.2) | 0.4 (1.2)

8. Secondary Outcome: Current Pain at Individual Time Points
Description: Current pain scores at the time of the data-collection phone call measured on a 0-10 Numeric Rating Scale with 0=no pain and 10=worst imaginable pain
Time Frame: Postoperative days 3 and 7; as well as Months 1 and 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation | Sham
Number analyzed (Participants) | 31 | 34
score on a scale
  Postoperative Day 3 | 0.4 (0.7) | 2.3 (2.3)
  Postoperative Day 7 | 0.3 (0.8) | 1.5 (2.2)
  Postoperative Month 1 | 0.3 (0.8) | 1.0 (1.8)
  Postoperative Month 4 | 0.1 (0.6) | 0.4 (0.9)

9. Secondary Outcome: Defense and Veterans Pain Rating Score
Description: Instrument designed to assess pain level specifically for active duty military and Veteran patient populations. It is a Likert scale from 0 (no pain) to 10 (worst imaginable pain).
Time Frame: Postoperative days 3, and 7; as well as Months 1 and 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peripheral Nerve Stimulation | Sham
Number analyzed (Participants) | 31 | 34
score on a scale
  Postoperative Day 3 | 1.4 (1.5) | 4.2 (2.3)
  Postoperative Day 7 | 1.1 (1.5) | 2.9 (2.5)
  Postoperative Month 1 | 1.3 (1.4) | 1.5 (2.0)
  Postoperative Month 4 | 0.6 (1.4) | 1.2 (1.7)

ADVERSE EVENTS:
Time Frame: 4 months following surgery
Arm/Group | Peripheral Nerve Stimulation | Sham
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/34
Other Adverse Events (participants affected / at risk) | 2/31 | 1/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peripheral Nerve Stimulation (N=31) | Sham (N=34)
Lead fracture during purposeful removal (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — The electrical lead fractured during purposeful removal. The remaining lead fragment is always left in situ and there were no adverse sequelae due to the fragments in the 4-month follow-up period.
Adhesive reaction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Erythema and irritation developed under the occlusive dressing holding the lead. The dressing and lead were removed and the erythema and irritation resolved without requiring treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT03481725/Prot_SAP_000.pdf